CLINICAL TRIAL: NCT04970667
Title: Clinical Study of Flupentixol and Melitracen Tablets in the Treatment of Non Random Emotional Disorder
Brief Title: Flupentixol and Melitracen Tablets in the Treatment of Emotional Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2017013
Record Dates: First submitted 2021-06-27; First posted 2021-07-21 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-06

CONDITIONS: Emotional Disorder; Neurologic Disorder
MeSH Terms: conditions — Nervous System Diseases | interventions — flupentixol, melitracen drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Flupentixol melitracen tablets (Experimental): The patients were treated with Flupentixol melitracen tablets according to their own conditions
  Interventions: Drug: Flupentixol melitracen tablets

INTERVENTIONS:
Drug: Flupentixol melitracen tablets — Patients were treated with Flupentixol and melitracen tablets for 12 weeks

SUMMARY:
To evaluate the efficacy and safety of Flupentixol melitracen tablets in the treatment of different types of non random emotional disorders

DETAILED DESCRIPTION:
Involuntary emotional expression disorder (ieed) is a kind of disorder of emotion control. Its main clinical feature is frequent short and violent uncontrollable crying and (or) laughing, which is different from mood disorder and self emotional expression.

The mixture of Flupentixol and melitracen is used for antidepressant. Melitracen is a tricyclic antidepressant, while Flupentixol is a neurodepressant in structure, but its dose in Deanxit has antidepressant properties.

The active components of Deanxit are Flupentixol dihydrochloride (Flupentixol) and melitracen (melitracen). Flupentixol is a thiazolyl (thioanthracene) antipsychotic, and melitracen is a tricyclic antidepressant. Low dose Flupentixol (0.5mg-3mg) has antidepressant and antianxiety effects, while melitracen has antidepressant effect. The mixture of the two components is used to treat mild to moderate mental disorders.

The purpose of this study was to evaluate the efficacy and safety of Flupentixol melitracen tablets in the treatment of different types of non random emotional disorders.

ELIGIBILITY:
Inclusion Criteria:

1. men and women aged 18-70;
2. Patients with nervous system diseases (such as stroke, amyotrophic lateral sclerosis, brain trauma, multiple sclerosis, Alzheimer's disease, etc.) accompanied by non random emotional expression disorder;
3. The informed consent form signed by the subject indicates that the subject has been informed of all the contents related to the study;
4. The subjects are willing and able to comply with the study visit schedule, treatment plan, laboratory examination and other study procedures.

Exclusion Criteria:

1. patients with acute infection, acute trauma, perioperative period and acute attack of chronic diseases;
2. Patients in critical condition or dying can not participate in this study;
3. Pregnant or lactating women;
4. Substance abuse patients;
5. Allergic to Deanxit;
6. Mental disorder; Coma;
7. Untreated angle closure glaucoma;
8. In the early recovery of myocardial infarction, patients with different degrees of heart block or arrhythmia and coronary artery ischemia;
9. Monoamine oxidase inhibitors were used;
10. Participated in any other studies involving studies or post marketing drugs within 30 days prior to screening;
11. According to the judgment of the researcher, there are other serious acute or chronic medical or psychiatric conditions or laboratory abnormalities that may increase the risks associated with participating in the trial or using the research products, or may affect the interpretation of the research results, which may make the subjects unsuitable for participating in the trial;
12. Inability and / or unwillingness to understand and / or comply with the protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of Flupentixol and Melitracen Tablets | The change of frequence of forced crying betwen baseline and twelfth week.
  Indicators of drug effectiveness: the difference between the number of crying episodes after 12 weeks of medication minus the number of crying episodes at baseline divided by the number of crying episodes at baseline. Complete remission was achieved when the attack disappeared, effective when the attack frequency decreased more than 50%, invalid when the attack frequency decreased less than or equal to 50%.

SECONDARY OUTCOMES:
Status of depression | At 12th week
  Status of depression was evaluated by Hamilton Depression Scale(HAMD),ranging from 0-54,the higher score means the worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Dongsheng Fan, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijin, China

IPD SHARING:
Plan to Share IPD: No